CLINICAL TRIAL: NCT01063101
Title: A Phase 1 Study to Evaluate the Effects of BAX 513 on Hemostatic Parameters in Healthy Volunteers
Brief Title: Phase 1 Dosing Study of BAX 513 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 950901
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — fucoidan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAX 513 (Experimental): Capsule - one of 5 dose levels (per randomization) - BID (= twice a day)
  Interventions: Other: Fucoidan (extract of Laminaria japonica)
- Capsule (cellulose) (Placebo Comparator): Capsule - one of 5 dose levels (per randomization) - BID
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fucoidan (extract of Laminaria japonica) — Capsule (300 mg/capsule) - oral administration - 5 different dose levels - BID
  Other Names: BAX 513
  Arms: BAX 513
Other: Placebo — Cellulose filled capsule - oral administration - 5 different dose levels - BID
  Arms: Capsule (cellulose)

SUMMARY:
The purpose of the study is to investigate whether orally administered BAX 513 (different doses administered for 5 days) affects hemostatic parameters in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Is >= 18 and < 70 years old at the time of screening
* Is able to provide signed and dated informed consent
* Is a healthy male or female adult
* If female and of childbearing potential, subject demonstrates a negative serum pregnancy test, and agrees to employ adequate birth control measures; (e.g., oral contraceptives, barrier method) for the duration of the study
* If female and receiving hormone replacement therapy (HRT), subject agrees to abstain from HRT for the duration of the study
* Subject's medical history and physical exam are normal
* Subject's lab values for complete blood count (CBC) and clinical chemistry are within normal ranges
* Is able to comprehend and comply with all aspects of the protocol and signed informed consent

Exclusion Criteria:

* If female, subject is pregnant or lactating at the time of study enrollment
* Has participated in another clinical study involving an investigational product (IP) or device within 30 days of screening or is scheduled to participate in another clinical study involving an IP or device during the course of this study
* Has a history of drug allergy in general or hypersensitivity to fucoidan containing products/foods or seafoods
* Medical and/or family history of thrombophilic tendencies, eg Protein C or S-deficiency, ATIII deficiency, FV Leiden mutation, Prothrombin 20210A mutation, lupus type inhibitor, antiphospholipid antibodies
* Medical history or clinical findings of a significant bleeding disorder
* Medical history of thrombotic events such as venous thromboembolism (VTE), myocardial infarction (MI), stroke or transient ischemic attack (TIA)
* Any other clinically relevant history of disease, eg malabsorption disorders, malignancies
* Any clinically significant abnormal laboratory values or abnormal ECG findings that in the opinion of the investigator are considered clinically relevant
* Seropositivity for HBs-Ag, HCV, HIV-1 or HIV-2 antibodies
* Symptoms of a clinically relevant illness within 3 weeks before screening
* A history of, or suspected, drug or alcohol abuse, or subject tests positive on a Drugs of Abuse screen within 1 week of dosing
* Intake of IP or related (fucoidan-containing) product within 1 week prior to study enrollment
* Any planned surgical or dental procedure during the course of this study
* Any recent surgery within 30 days of enrollment
* Presence of signs or symptoms consistent with an infection, such as fever, chills, or nausea during screening in this study
* Chronic or regular use of aspirin, ibuprofen, coumarin derivatives, antiplatelet drugs, within 1 week before enrollment
* Use of concomitant drugs diclofenac or [paracetamol if > 2 g/day] within 1 week before first day of study dosing
* Plasmapheresis or platelet donation within 3 weeks of screening and until final visit
* Any medical condition that may compromise the ability to give written informed consent or to comply with the study protocol
* Subject is a member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01-29 (Actual); Primary Completion 2010-07-22 (Actual); Study Completion 2010-08-01 (Actual)

PRIMARY OUTCOMES:
Change in peak thrombin concentration from baseline as measured by the Thrombin Generation Assay (TGA). | 7 months (= anticipated study duration)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- University Clinic for Clinical Pharmacology, General Hospital Vienna, Vienna, Austria